CLINICAL TRIAL: NCT04308031
Title: Efficacy of Ivabradine as a Treatment Modality for Both Rate Control and Heart Failure Medication in Patient With Both Persistent Atrial Fibrillation and Heart Failure With Reduce and Mid-range Ejection Fraction
Brief Title: Efficacy of Ivabradine in Patient With Both Persistent Atrial Fibrillation and Heart Failure With Reduce Ejection Fraction
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chun-Yao Huang (Other)
Responsible Party: Sponsor-Investigator, Chun-Yao Huang, Attending physician, Taipei Medical University Hospital
Organization: Taipei Medical University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N201801089
Record Dates: First submitted 2019-05-09; First posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Atrial Fibrillation; Ivabradine; Heart Failure
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure | interventions — Ivabradine; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ivabradine (Experimental): Subject will be randomly assigned to either Ivabradine or Digoxin group. Ivabradine starting dose is 2.5 mg twice daily(BID). ECG will be performed at each visit during the treatment phase and dose will be adjusted based on the heart rate result from the ECG. Total treatment phase is 16 weeks ( 4 months).
  Interventions: Drug: Ivabradine 5 mg [Corlanor]
- Digoxin (Active Comparator): Subject will be randomly assigned to either Ivabradine or Digoxin group. Digoxin starting dose is 0.125mg once daily(QD) in estimated Glomerular filtration rate(eGFR)>60， 0.125mg every other day (QOD) in estimated Glomerular filtration rate(eGFR)<60. Dose adjustment will be based on heart rate result from ECG performed at each treatment visit and Digoxin level from blood sample collected from each visit during treatment phase. Total treatment phase is 16 weeks ( 4 months).
  Interventions: Drug: Digoxin 0.25 mg

INTERVENTIONS:
Drug: Ivabradine 5 mg [Corlanor] — Starting dose: Ivabradine 2.5mg twice daily (BID) Max Dose: Ivabradine 7.5 mg twice daily (BID)
  Arms: Ivabradine
Drug: Digoxin 0.25 mg — Starting dose: 0.125mg once daily (QD) in estimated Glomerular filtration rate(eGFR)>60， 0.125mg once every other day (QOD) in estimated Glomerular filtration rate(eGFR)<60 Max dose: 0.25 once daily (QD)
  Arms: Digoxin

SUMMARY:
Atrial fibrillation (AF) is the most common arrhythmia encountered in clinical practice. Previous studies have shown that rate control strategy in AF is non-inferior to rhythm control strategy, in terms of stroke and mortality risk. In addition, rate control strategy is associated with lower risk of hospitalization and non-cardiovascular mortality. Therefore, rate control is an essential strategy to improve quality of life, decrease morbidity and prevent tachycardia-induced cardiomyopathy in AF patients. The recommended rate control agents include beta-blocker, nondihydropyridine calcium-channel blocker (CCB), digoxin and amiodarone. However, in heart failure with reduced ejection fraction patient, the medication of rate control were beta-blocker than digoxin. But several clinical observation study show excess mortality in AF patients. Ivabradine, a If inhibitor, it is well-established that a pacemaker current, If current, is functionally expressed in the sinus node . Previous studies have shown that Ivabradine, If inhibitor, significantly reduces sinus rate and improves prognosis in patients with systolic heart failure. Interestingly, several investigators found that hyperpolarization- activated cyclic nucleotidylated channel 4 current (HCN4), the main isoform of the channel responsible for If current, is also functionally expressed in the Atrioventricular node(AV node). Recent data have shown that inhibition of If current slows AV node conduction in animals and humans. Thus, we want to compare the effect of Ivabradine on ventricular rate with digoxin in this study.

ELIGIBILITY:
Inclusion Criteria:

1. The patient with persistent or permanent atrial fibrillation(24hr ECG) with HFrEF and HFmrEF.
2. After maximal tolerance dose beta-blocker(Bisoprolol 20mg/day，Carvedilol 50mg/day) or intolerant to beta-blocker the resting heart rate from ECG is still faster than 100 or resting heart rate from ECG is greater than 80 but still with symptoms of short of breath and palpitation.
3. Stable heart rhythm medication.(no change of medication in recently one week)
4. Age 20 to 90 years old.
5. The subject must be an adult who can read himself/herself and walk independently.

Exclusion Criteria:

1. Used medication with interaction with digoxin : Clarithromycin, Erythromycin, Azithromycin, ritonavir, lopinavir/ritonavir, Doxycycline, Minocycline, tetracycline。
2. Used medication with interaction with ivabradine: voriconazole, posaconazole, fluconazole, Ombitasvir, Dasabuvir, Carbamazepine, Enzalutamide, Fosphenytoin, Mitotane, Phenobarbital, Phenytoin, Rifampicin
3. Cardiogenic shock.
4. History of symptomatic bradycardia.
5. Renal insufficiency:eGFR<30 ml/min/1.73m2
6. Pregnancy
7. Heart failure due to congenital heart
8. Severe hypotension(<90/50mmHg)

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-08-26 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Heart rate change | 24 hr ECG test will be performed at Screening phase and End of Treatment visit(Visit5/Week 16).
  To compare Heart Rate change monitored from 24 hr ECG. Test will be performed at Baseline (screening phase, 4 weeks time between screening/Informed consent and Randomization visit) and treatment completion (Visit 5/Week 16). Total treatment phase is 16 weeks.
6 minute walk test change | Test will be performed at Randomization visit (V1/Week0) and treatment completion (Visit 5/Week 16).
  To compare 6 minute walking test walking distance change between Randomization visit(Visit 1/Week 0) and treatment completion(Visit 5/Week 16). Total Treatment phase is 16 weeks.
N-terminal pro-brain natriuretic peptide(NT-Pro BNP) change | Blood sample will be collected at Screening phase and End of Treatment visit(Visit5/Week 16).
  To compare NT-Pro BNP change from blood sample collected at Baseline (screening phase, 4 weeks time between screening/informed consent and Randomization visit) and treatment completion (Visit 5/Week 16). Total treatment phase is 16 weeks.
1-10 Borg Rating of Perceived Exertion Scale change | Borg's score will be tested at Randomization visit (V1/Week0) and treatment completion (Visit 5/Week 16).
  To compare 1-10 Borg Rating of Perceived Exertion Scale change between Randomization visit (Visit1/Week0) and treatment completion (Visit 5/Week 16). Total Treatment phase is 16 weeks. The number 1-10 Borg Rating of Perceived Exertion Scale will be obtained pre and post 6 minutes walk test. The value of 1-10 Borg Rating of Perceived Exertion Scale pre 6 minutes walking test will be compared between Randomization visit (Visit1/Week0) and treatment completion (Visit 5/Week 16), and the same type of comparison will be performed for 1-10 Borg Rating of Perceived Exertion Scale values post 6 minute walk test. Rating score is as below: 0=Rest, 1=really easy, 2=easy, 3=moderate, 4=sort of hard, 5=hard, 6= between 5 and 7, 7=really hard, 8=between 7 and 9, 9=really really hard, 10=Maximal: just like my hardest race. Decrease in score value compared between Randomization visit (Visit1/Week0) and treatment completion (Visit 5/Week 16) represents better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No